CLINICAL TRIAL: NCT01934881
Title: Voltage Only Adjustment Versus Multiple Parameters Adjustment of Bilateral Subthalamic Deep Brain Stimulation Treatment in Parkinson's Disease Patients: a Protocol of a Prospective, Multicenter, and Observational Study.
Brief Title: Voltage Only Adjustment Versus Multiple Parameters Adjustment of Bilateral STN DBS Treatment in PD Patients.
Acronym: VOMPDS
Status: Completed | Type: Observational
Sponsor: Chen Ling (Other)
Collaborators: Prince of Wales Hospital, Shatin, Hong Kong (Other); Shenzhen Second People's Hospital (Other)
Responsible Party: Sponsor-Investigator, Chen Ling, MD,PhD, First Affiliated Hospital, Sun Yat-Sen University
Organization: First Affiliated Hospital, Sun Yat-Sen University (Other)
Other Study IDs: [2013] 19
Record Dates: First submitted 2013-08-30; First posted 2013-09-04 (Estimated); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Parkinson's Disease
Keywords: Deep Brain Stimulation; programming
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (2):
- group I: Voltage adjustment only
  Interventions: Device: voltage adjustment only
- group II: Multiple parameters adjustment
  Interventions: Device: Multiple parameters adjustment

INTERVENTIONS:
Device: voltage adjustment only — Only voltage will be adjusted in all programming sections.
  Groups: group I
Device: Multiple parameters adjustment — More than one parameter, including voltage, frequency and pulse width, will be adjusted in the programming sections.
  Groups: group II

SUMMARY:
The programming of subthalamic nucleus (STN) deep brain stimulation (DBS) for Parkinson's disease (PD) is complex work because the parameter setting has not been standardized so far. The objective of the present study is to set up a standardized programming algorithm for Chinese PD patients treated with bilateral STN DBS.

DETAILED DESCRIPTION:
A total of 150 subjects will be recruited from the concurrent NCT01922388 study and followed up for four years. All patients will be evaluated using the Movement Disorder Society-sponsored revision of the Unified Parkinson's Disease Rating Scale (MDS-UPDRS) part III at baseline (one week before surgery) and at 12 and 48 months postoperatively.

Stimulation parameters setting: The first programming is performed at 4 weeks after surgery. Bilateral contacts are as cathode for monopolar configuration. The initial voltage, pulse width and frequency are bilaterally 1.0-1.5 V, 60 μs and 130 Hz for each individual, respectively. Voltage is gradually increased to a stable level first, until the optimal efficacy is achieved. Two weeks later, when patients came back to hospital for reprogramming, the voltage is also first adjusted to optimize the stimulation parameters. Either pulse width or frequency will be adjusted when increasing voltage more than 0.4 V for one time still can not get satisfactory outcomes. The frequency is adjusted when bilateral symptoms are unresponsive to voltage. Frequency is increased by 15-20 Hz for each time. Pulse width is then adjusted for the satisfactory clinical response of unilateral symptoms which are not satisfied after increasing voltage or frequency. Pulse width is increased to 90 μs if necessary (e.g. severe tremor).

Groups: Patients are divided into two groups according to the parameter settings during follow-up. Group I: patients with voltage adjustment only. The pulse width is kept to 60 μs and frequency to 130 Hz constant throughout the follow-up period. Group II: patients with adjustment of more than two stimulation parameters (voltage, pulse width or frequency) during the follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. The patients with the idiopathic Parkinson's disease with good response to levodopa medication (i.e. more than 30% improvement in the MDS-UPDRS Part III score of the motor function examination(Goetz et al., 2008b) after an acute levodopa medication challenge);
2. Disease duration ≥4 years;
3. The patients with the fluctuations and/or dyskinesias;
4. The patients with age ranging from 18 to 75 years old;
5. The patients with normal brain on the MRI;
6. The patients with the absence of dementia (Mini-Mental State Examination scores of≥ 26) ;
7. The patients with the absence of severe psychiatric diseases;
8. The patients who provided the written informed consent

Exclusion Criteria:

1. The patients with severe metabolic diseases;
2. The patients with severe cardiac/respiratory/renal/hepatic diseases;
3. The patients having secondary parkinsonism or multiple system atrophies;
4. The patients who illiterate or having insufficient language skills to complete the questionnaires;
5. The patients who had poor compliance and unreasonable expectation;
6. Women who were pregnant or breast feeding;
7. The patients with the simultaneous participation in another clinical trial

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: PD Patients are selected from the outpatient department of three centres.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2013-09 (Actual); Primary Completion 2022-12 (Actual); Study Completion 2022-12 (Actual)

PRIMARY OUTCOMES:
Changes in motor symptoms (tremor, rigidity, bradykinesia and postural stability) evaluated by MDS-UPDRS Part III in off medication /on stimulation state | From baseline to 12 and 48 months
  Motor subscores

SECONDARY OUTCOMES:
Changes in 39-item Parkinson's Disease Questionnaire (PDQ-39) scores | From baseline to 12 and 48 months
  Quality of life
Changes in levodopa equivalent daily dosage (LEDD) | From baseline to 12 and 48 months
  Medication dosage

CONTACTS AND LOCATIONS:
Overall Officials: Ling Chen, MD, PhD, Principal Investigator — First Affiliated Hospital, Sun Yat-Sen University
Locations (1):
- the First Affiliated Hospital, Sun Yat-sen University, Guangzhou, Guangdong, China

REFERENCES:
- [Derived] Xu SH, Yang C, Xian WB, Gu J, Liu JL, Jiang LL, Ye J, Liu YM, Guo QY, Zheng YF, Wu L, Chen WR, Pei Z, Chen L. Voltage adjustment improves rigidity and tremor in Parkinson's disease patients receiving deep brain stimulation. Neural Regen Res. 2018 Feb;13(2):347-352. doi: 10.4103/1673-5374.226406. PMID 29557387